CLINICAL TRIAL: NCT02559427
Title: Impact of 3-week SPA Therapy on Sleep Apnea in Patients With Obstructive Sleep Apnea Syndrome and Chronic Venous Insufficiency: A Randomized, Controlled Study
Brief Title: SPA Therapy in the Treatment of Sleep Apnea Syndrome
Acronym: THERMA-SAS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients randomized after more than one year sponsor decided to withdrawn the study.
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: Floralis (Industry); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THERMA SAS
Record Dates: First submitted 2015-07-29; First posted 2015-09-24 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Obstructive Sleep Apnea Syndrome; Chronic Venous Insufficiency
Keywords: sleep apnea; Venous Insufficiency; SPA treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate SPA treatment (Active Comparator): 3-week immediate SPA treatment (soon after randomization)
  Interventions: Other: 3-week immediate SPA treatment
- Late SPA treatment (Sham Comparator): 3-week late SPA treatment (soon after primary endpoint at 4 1/2 months visit)
  Interventions: Other: 3-week late SPA treatment

INTERVENTIONS:
Other: 3-week immediate SPA treatment — a comprehensive program soon after randomization including sessions of balneotherapy, diet information, exercise training. The most adapted to the concerned pathology and common to all SPA resorts (walk in a specially pool, whirlpool bath with automatic air and water massages cycles, massages shower...)
  Other Names: Immediate SPA treatment
  Arms: Immediate SPA treatment
Other: 3-week late SPA treatment — a comprehensive program after 4.5 months, including sessions of balneotherapy, diet information, exercise training. The most adapted to the concerned pathology and common to all SPA resorts (walk in a specially pool, whirlpool bath with automatic air and water massages cycles, massages shower...)
  Other Names: Late SPA treatment
  Arms: Late SPA treatment

SUMMARY:
The purpose of this study is to determine whether 3-week of SPA therapy improves sleep apnea in patients with chronic venous insufficiency and concomitant Obstructive Sleep Apnea Syndrome (OSAS).

DETAILED DESCRIPTION:
Obstructive Sleep Apnea Syndrome (OSAS), characterized by repetitive episodes of partial or complete upper airway (UA) obstruction, is highly prevalent in the general population (2% in women, 4% in men). OSAS is associated with hypersomnolence and it increases the risk of cardiovascular morbidity and mortality. Its pathogenesis is largely multifactorial. In patients with chronic venous insufficiency, fluid retention contributes to this pathogenesis: during the day, fluid accumulates in the legs due to gravity ; during sleep in recumbent position, this accumulated fluid redistributes rostrally in the neck and causes upper airway narrowing and predisposes to OSAS.

The hypothesis is that a comprehensive treatment program for chronic venous insufficiency (SPA therapy) would reduce sleep apnea in patients with chronic venous insufficiency and concomitant sleep apnea Syndrome.

The objective is to assess the efficacy of a 3-week SPA therapy on attenuation of sleep apnea in this population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Chronic Venous Insufficiency with oedema (CEAP clinical classes C3 to C5) and concomitant Sleep Apnea Syndrome (AHI > 15 events/hour)
* Patient in stable state (no change in medical treatment and no hospitalization for respiratory, cardiac or metabolic event in the 2 months preceding inclusion)
* Patient available for a program of 3-week SPA Therapy

Exclusion Criteria:

* Patient with no social insurance
* Pregnant and nursing woman
* Patient detained by judicial order
* Patient with contra-indication to SPA therapy
* Patient with chronic venous insufficiency < CEAP C3 or CEAP C6
* Patient already treated by class IV compression stockings for severe veinolymphatic insufficiency
* Patient already treated for sleep apnea
* Patient who have already benefited of SPA therapy (any type) within 9 months before the enrollment
* Patient with severe comorbidities
* Patient who could not respect the constraints related to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 4.5 months
  Variation in AHI according to the allocation group

SECONDARY OUTCOMES:
Specific Quality of life | 4.5 months
  Variation in the scores of CIVIQ 20 according to the allocation group (Specific quality of life scale for venous insufficiency)
Global Quality of life | 4.5 months
  Variation in the score of EUROQUOL according to the allocation group (Global quality of life scale)
severity of sleep apnea | 4.5 months
  Variation of AHI according to the severity of sleep apnea at inclusion. Moderate sleep apnea (AHI <30) vs Severe Sleep apnea (AHI >30) at inclusion
Nocturnal hypoxemia | 4.5 months
  Nocturnal hypoxemia is assessed by mean SpO2 and time spent with SpO2<90%
Clinically significant improvement of OSAS | 4.5 months
  Clinically significant improvement is defined with a reduction in AHI by 50% or more and a reduction in oxygen desaturation index by 50% or more
Sleep duration | 4.5 months
  Mean sleep duration is assessed by actigraphy over a period of 7 days.
Quality of Sleep | 4.5 months
  Quality of sleep is assessed by Quebec Quality of life Questionnaire
Daytime sleepiness | 4.5 months
  Sleepiness is assessed by Epworth sleepiness scale
Variation of interstitial fluid | 4.5 months
  bioimpedance is used to measure interstitial fluid
Long term efficacy | 1 year
  Long term efficacy is measured by nocturnal respiratory polygraphy only in patients who are not treated by CPAP
Venous insufficiency classification | 1 year
  Variation of venous insufficiency is assessed by CEAP classification
Venous insufficiency variation | 1 year
  Variation of venous insufficiency is assessed by Villalta score
Venous insufficiency examination | 1 year
  Variation of venous insufficiency is assessed by leg circumferences
long term effect of the SPA treatment on primary outcome | 1 year
  confirmation of the long term effect of the SPA treatment at 1 year for the control group. Primary outcome evolution between 4.5 months and 12 months (evolution of AHI)
long term effect of the SPA treatment on specific quality of life | 1 year
  confirmation of the long term effect of the SPA treatment at 1 year for the control group. Evolution between 4.5 months and 12 months of specific quality of life with CIVIQ 20 scale
long term effect of the SPA treatment on global quality of life | 1 year
  confirmation of the long term effect of the SPA treatment at 1 year for the control group. Evolution between 4.5 months and 12 months of global quality of life with EUROQUOL Scale
long term effect of the SPA treatment on venous insufficiency | 1 year
  confirmation of the long term effect of the SPA treatment at 1 year for the control group. Evolution between 4.5 months and 12 months of venous insufficiency
long term effect of the SPA treatment on specific treatment of OSAS | 1 year
  confirmation of the long term effect of the SPA treatment at 1 year for the control group. Evolution between 4.5 months and 12 months. The long term effect will be confirmed if patients did not require a specific treatment of OSAS (for example CPAP (Continuous Positive Airway Pressure).
benefit for patients with first SPA treatment | 4.5 months
  stratification at randomization (first SPA treatment or not) to evaluate a higher benefit (variation of Apnea-Hypopnea Index (AHI)) for patients with first SPA treatment. Comparison of patients with first SPA treatment or not on primary outcome according to the allocation group.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis PEPIN, MD, Principal Investigator — University Hospital, Grenoble
Locations (8):
- France (8):
  - Medical pratice (angiology), Annecy
  - Medical practice (angiology), Bourgoin
  - Medical practice (angiology), Castelnau-le-Lez
  - University Hospital Grenoble, Grenoble
  - Medical pratice (angiology), Grenoble
  - Clinic Beau Soleil, Montpellier
  - Medical pratice (angiology), Tarbes
  - Medical practice (angiology), Valence

REFERENCES:
- [Background] Punjabi NM. The epidemiology of adult obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):136-43. doi: 10.1513/pats.200709-155MG. PMID 18250205
- [Background] Caffo B, Diener-West M, Punjabi NM, Samet J. A novel approach to prediction of mild obstructive sleep disordered breathing in a population-based sample: the Sleep Heart Health Study. Sleep. 2010 Dec;33(12):1641-8. doi: 10.1093/sleep/33.12.1641. PMID 21120126
- [Background] Young T, Palta M, Dempsey J, Peppard PE, Nieto FJ, Hla KM. Burden of sleep apnea: rationale, design, and major findings of the Wisconsin Sleep Cohort study. WMJ. 2009 Aug;108(5):246-9. PMID 19743755
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Monahan K, Storfer-Isser A, Mehra R, Shahar E, Mittleman M, Rottman J, Punjabi N, Sanders M, Quan SF, Resnick H, Redline S. Triggering of nocturnal arrhythmias by sleep-disordered breathing events. J Am Coll Cardiol. 2009 Nov 3;54(19):1797-804. doi: 10.1016/j.jacc.2009.06.038. PMID 19874994
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Teran-Santos J, Jimenez-Gomez A, Cordero-Guevara J. The association between sleep apnea and the risk of traffic accidents. Cooperative Group Burgos-Santander. N Engl J Med. 1999 Mar 18;340(11):847-51. doi: 10.1056/NEJM199903183401104. PMID 10080847
- [Background] Yaggi HK, Concato J, Kernan WN, Lichtman JH, Brass LM, Mohsenin V. Obstructive sleep apnea as a risk factor for stroke and death. N Engl J Med. 2005 Nov 10;353(19):2034-41. doi: 10.1056/NEJMoa043104. PMID 16282178
- [Background] Flemons WW, Reimer MA. Development of a disease-specific health-related quality of life questionnaire for sleep apnea. Am J Respir Crit Care Med. 1998 Aug;158(2):494-503. doi: 10.1164/ajrccm.158.2.9712036. PMID 9700127
- [Background] Dempsey JA, Veasey SC, Morgan BJ, O'Donnell CP. Pathophysiology of sleep apnea. Physiol Rev. 2010 Jan;90(1):47-112. doi: 10.1152/physrev.00043.2008. PMID 20086074
- [Background] Levy P, Pepin JL, Dematteis M. Pharyngeal neuropathy in obstructive sleep apnea: where are we going? Am J Respir Crit Care Med. 2012 Feb 1;185(3):241-3. doi: 10.1164/rccm.201111-1992ED. No abstract available. PMID 22298363
- [Background] Javaheri S. Sleep disorders in systolic heart failure: a prospective study of 100 male patients. The final report. Int J Cardiol. 2006 Jan 4;106(1):21-8. doi: 10.1016/j.ijcard.2004.12.068. PMID 16321661
- [Background] Yumino D, Wang H, Floras JS, Newton GE, Mak S, Ruttanaumpawan P, Parker JD, Bradley TD. Prevalence and physiological predictors of sleep apnea in patients with heart failure and systolic dysfunction. J Card Fail. 2009 May;15(4):279-85. doi: 10.1016/j.cardfail.2008.11.015. Epub 2009 Jan 21. PMID 19398074
- [Background] de Oliveira Rodrigues CJ, Marson O, Tufic S, Kohlmann O Jr, Guimaraes SM, Togeiro P, Ribeiro AB, Tavares A. Relationship among end-stage renal disease, hypertension, and sleep apnea in nondiabetic dialysis patients. Am J Hypertens. 2005 Feb;18(2 Pt 1):152-7. doi: 10.1016/j.amjhyper.2004.08.028. PMID 15752940
- [Background] Logan AG, Perlikowski SM, Mente A, Tisler A, Tkacova R, Niroumand M, Leung RS, Bradley TD. High prevalence of unrecognized sleep apnoea in drug-resistant hypertension. J Hypertens. 2001 Dec;19(12):2271-7. doi: 10.1097/00004872-200112000-00022. PMID 11725173
- [Background] Yumino D, Redolfi S, Ruttanaumpawan P, Su MC, Smith S, Newton GE, Mak S, Bradley TD. Nocturnal rostral fluid shift: a unifying concept for the pathogenesis of obstructive and central sleep apnea in men with heart failure. Circulation. 2010 Apr 13;121(14):1598-605. doi: 10.1161/CIRCULATIONAHA.109.902452. Epub 2010 Mar 29. PMID 20351237
- [Background] Friedman O, Bradley TD, Chan CT, Parkes R, Logan AG. Relationship between overnight rostral fluid shift and obstructive sleep apnea in drug-resistant hypertension. Hypertension. 2010 Dec;56(6):1077-82. doi: 10.1161/HYPERTENSIONAHA.110.154427. Epub 2010 Nov 8. PMID 21060007
- [Background] Elias RM, Bradley TD, Kasai T, Motwani SS, Chan CT. Rostral overnight fluid shift in end-stage renal disease: relationship with obstructive sleep apnea. Nephrol Dial Transplant. 2012 Apr;27(4):1569-73. doi: 10.1093/ndt/gfr605. Epub 2011 Nov 5. PMID 22058175
- [Background] Redolfi S, Arnulf I, Pottier M, Lajou J, Koskas I, Bradley TD, Similowski T. Attenuation of obstructive sleep apnea by compression stockings in subjects with venous insufficiency. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1062-6. doi: 10.1164/rccm.201102-0350OC. PMID 21836140
- [Background] Rapoport DM, Garay SM, Epstein H, Goldring RM. Hypercapnia in the obstructive sleep apnea syndrome. A reevaluation of the "Pickwickian syndrome". Chest. 1986 May;89(5):627-35. doi: 10.1378/chest.89.5.627. PMID 3516586
- [Background] Sullivan CE, Issa FG, Berthon-Jones M, Eves L. Reversal of obstructive sleep apnoea by continuous positive airway pressure applied through the nares. Lancet. 1981 Apr 18;1(8225):862-5. doi: 10.1016/s0140-6736(81)92140-1. PMID 6112294
- [Background] Giles TL, Lasserson TJ, Smith BH, White J, Wright J, Cates CJ. Continuous positive airways pressure for obstructive sleep apnoea in adults. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD001106. doi: 10.1002/14651858.CD001106.pub3. PMID 16855960
- [Background] Haentjens P, Van Meerhaeghe A, Moscariello A, De Weerdt S, Poppe K, Dupont A, Velkeniers B. The impact of continuous positive airway pressure on blood pressure in patients with obstructive sleep apnea syndrome: evidence from a meta-analysis of placebo-controlled randomized trials. Arch Intern Med. 2007 Apr 23;167(8):757-64. doi: 10.1001/archinte.167.8.757. PMID 17452537
- [Background] Marin JM, Agusti A, Villar I, Forner M, Nieto D, Carrizo SJ, Barbe F, Vicente E, Wei Y, Nieto FJ, Jelic S. Association between treated and untreated obstructive sleep apnea and risk of hypertension. JAMA. 2012 May 23;307(20):2169-76. doi: 10.1001/jama.2012.3418. PMID 22618924
- [Background] Sharma SK, Agrawal S, Damodaran D, Sreenivas V, Kadhiravan T, Lakshmy R, Jagia P, Kumar A. CPAP for the metabolic syndrome in patients with obstructive sleep apnea. N Engl J Med. 2011 Dec 15;365(24):2277-86. doi: 10.1056/NEJMoa1103944. PMID 22168642 (Retraction: PMID 24171540 Sharma SK, Agrawal S, Damodaran D, Sreenivas V, Kadhiravan T, Lakshmy R, Jagia P, Kumar A. N Engl J Med. 2013 Oct 31;369(18):1770)
- [Background] Papandreou C, Schiza SE, Bouloukaki I, Hatzis CM, Kafatos AG, Siafakas NM, Tzanakis NE. Effect of Mediterranean diet versus prudent diet combined with physical activity on OSAS: a randomised trial. Eur Respir J. 2012 Jun;39(6):1398-404. doi: 10.1183/09031936.00103411. Epub 2011 Oct 27. PMID 22034645
- [Background] Kline CE, Crowley EP, Ewing GB, Burch JB, Blair SN, Durstine JL, Davis JM, Youngstedt SD. The effect of exercise training on obstructive sleep apnea and sleep quality: a randomized controlled trial. Sleep. 2011 Dec 1;34(12):1631-40. doi: 10.5665/sleep.1422. PMID 22131599
- [Background] Mirrakhimov AE. Physical exercise related improvement in obstructive sleep apnea. Look for the rostral fluid shift. Med Hypotheses. 2013 Feb;80(2):125-8. doi: 10.1016/j.mehy.2012.11.007. Epub 2012 Dec 3. PMID 23218530
- [Background] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131
- [Background] Gottlieb DJ, Yenokyan G, Newman AB, O'Connor GT, Punjabi NM, Quan SF, Redline S, Resnick HE, Tong EK, Diener-West M, Shahar E. Prospective study of obstructive sleep apnea and incident coronary heart disease and heart failure: the sleep heart health study. Circulation. 2010 Jul 27;122(4):352-60. doi: 10.1161/CIRCULATIONAHA.109.901801. Epub 2010 Jul 12. PMID 20625114
- [Background] Strollo PJ Jr, Soose RJ, Maurer JT, de Vries N, Cornelius J, Froymovich O, Hanson RD, Padhya TA, Steward DL, Gillespie MB, Woodson BT, Van de Heyning PH, Goetting MG, Vanderveken OM, Feldman N, Knaack L, Strohl KP; STAR Trial Group. Upper-airway stimulation for obstructive sleep apnea. N Engl J Med. 2014 Jan 9;370(2):139-49. doi: 10.1056/NEJMoa1308659. PMID 24401051
- [Background] Chan AS, Sutherland K, Schwab RJ, Zeng B, Petocz P, Lee RW, Darendeliler MA, Cistulli PA. The effect of mandibular advancement on upper airway structure in obstructive sleep apnoea. Thorax. 2010 Aug;65(8):726-32. doi: 10.1136/thx.2009.131094. PMID 20685749
- [Background] Vickers AJ, Altman DG. Statistics notes: Analysing controlled trials with baseline and follow up measurements. BMJ. 2001 Nov 10;323(7321):1123-4. doi: 10.1136/bmj.323.7321.1123. No abstract available. PMID 11701584
- [Background] Kahn SR, Partsch H, Vedantham S, Prandoni P, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of post-thrombotic syndrome of the leg for use in clinical investigations: a recommendation for standardization. J Thromb Haemost. 2009 May;7(5):879-83. doi: 10.1111/j.1538-7836.2009.03294.x. Epub 2009 Jan 19. PMID 19175497